CLINICAL TRIAL: NCT03060135
Title: Comparing the Efficacy of Several Popular Online Interventions to Reduce Hazardous Alcohol Consumption: Randomized Controlled Trial
Brief Title: Comparing the Efficacy of Several Popular Online Interventions to Reduce Hazardous Alcohol Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11/13/2016
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Intervention: Control (No Intervention): A questionnaire that asks individuals what components of an online intervention they might find useful.
- Check Your Drinking (CYD) (Active Comparator): The CYD is a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Interventions: Behavioral: Check Your Drinking
- Hello Sunday Morning (Experimental): Internet based program designed to assess drinking patterns, and support self-determined goals for abstinence, by providing users with an online platform and community to discuss progress and goals.
  Interventions: Behavioral: Hello Sunday Morning

INTERVENTIONS:
Behavioral: Check Your Drinking — A anonymous brief survey designed to provide normative feedback of individual's drinking with the intent of motivating reductions in drinking
  Arms: Check Your Drinking (CYD)
Behavioral: Hello Sunday Morning — Brief online intervention that allows Individual's reflect on their drinking reductions progress and goals.
  Arms: Hello Sunday Morning

SUMMARY:
There are a number of popular, freely available online interventions targeting hazardous alcohol consumption. Unfortunately, most have limited or no published evidence regarding their efficacy. Of particular interest is the intervention, 'Hello Sunday Morning.' The current project proposes to evaluate its' efficacy employing a RCT, using The Check Your Drinking intervention as an active comparator in the trial.

Participants will be recruited through Amazon's MTurk crowdsourcing platform. Potential participants identified as problem drinkers based on an initial survey will be invited to complete another survey in 6 months time. Those who agree to be followed-up will be assigned by chance to be asked versus not asked to access one of the interventions and then recontacted 6 months later to ask about their drinking and their impressions of the online intervention. The primary hypothesis to be tested is that participants receiving access to any of the online interventions will report a greater level of reduction in number of drinks in a typical week between the baseline survey and six-month follow-up as compared to participants in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* A score of 8 or over on the Alcohol Use Disorders Identification Test (AUDIT)
* Typically consumes 15 or more drinks per week,
* Willingness to complete a 6-month follow-up survey

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Change in the variable, number of drinks in a typical week, from baseline measurement to 6-month follow-up | 6 months
  Sum of number of drinks consumed in a typical week

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schell C, Godinho A, Cunningham JA. To thine own self, be true: Examining change in self-reported alcohol measures over time as related to socially desirable responding bias among people with unhealthy alcohol use. Subst Abus. 2021;42(1):87-93. doi: 10.1080/08897077.2019.1697998. Epub 2020 Feb 10. PMID 32040383
- [Derived] Cunningham JA, Godinho A, Bertholet N. Outcomes of two randomized controlled trials, employing participants recruited through Mechanical Turk, of Internet interventions targeting unhealthy alcohol use. BMC Med Res Methodol. 2019 Jun 14;19(1):124. doi: 10.1186/s12874-019-0770-4. PMID 31200648
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research